CLINICAL TRIAL: NCT00482079
Title: A Multicenter, Double-Blind, Randomized, Placebo- and Active-Controlled Dose-Range Finding Study of MK0431 in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: A Study of MK0431 in Patients With Type 2 Diabetes (0431-010)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0431-010; 2007_578
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: MK0431, sitagliptin phosphate / Duration of Treatment: 21 Weeks
Drug: Comparator: placebo (unspecified) / Duration of Treatment: 21 Weeks

SUMMARY:
A dose-ranging study of MK0431 in patients with type 2 diabetes who have inadequate control of their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 70, You are a man or non-pregnant woman

Exclusion Criteria:

* Have a history of type I diabetes
* You are on a weight loss program with ongoing weight loss or taking weight loss medications
* You have a history of minor surgery
* You have received investigational drugs within 8 weeks of study start
* You have hepatitis B or C

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2003-05-13 (Actual); Primary Completion 2004-08-25 (Actual); Study Completion 2006-06-15 (Actual)

PRIMARY OUTCOMES:
To asses the effectiveness of MK0431 compared to placebo | over 12 weeks

SECONDARY OUTCOMES:
To test the safety and tolerability of MK0431 in patients with type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Scott R, Wu M, Sanchez M, Stein P. Efficacy and tolerability of the dipeptidyl peptidase-4 inhibitor sitagliptin as monotherapy over 12 weeks in patients with type 2 diabetes. Int J Clin Pract. 2007 Jan;61(1):171-80. doi: 10.1111/j.1742-1241.2006.01246.x. Epub 2006 Dec 5. PMID 17156104
- [Derived] Ommen ES, Xu L, O'Neill EA, Goldstein BJ, Kaufman KD, Engel SS. Comparison of treatment with sitagliptin or sulfonylurea in patients with type 2 diabetes mellitus and mild renal impairment: a post hoc analysis of clinical trials. Diabetes Ther. 2015 Mar;6(1):29-40. doi: 10.1007/s13300-015-0098-y. Epub 2015 Jan 30. PMID 25633134
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html